CLINICAL TRIAL: NCT00858416
Title: Efficacy of Combined Local Mechanical Vibrations, Continuous Passive Motion and Thermotherapy in the Management of Osteoarthritis of the Knee
Brief Title: Combined Vibrations, Passive Motion and Thermotherapy for Knee Osteoarthritis
Acronym: KC-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kineticure (Industry)
Responsible Party: Dr. Garry S Kitay, Jacksonville Orthopedic Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KC-01
Record Dates: First submitted 2009-03-02; First posted 2009-03-09 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis; Knee Pain
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AB (Experimental): First active then Sham
  Interventions: Device: "Kineticure System" followed by sham
- BA (Sham Comparator): First sham then active
  Interventions: Device: sham followed by "Kineticure System"

INTERVENTIONS:
Device: "Kineticure System" followed by sham — 20 minutes sessions with knee brace (integrated heating pad, a vibration unit and a foot pedal that delivers continuous passive motion) during the first 4 weeks followed by 2 weeks wash out and 4 weeks of sham device
  Other Names: Kineticure System
  Arms: AB
Device: sham followed by "Kineticure System" — sham device during the first 4 weeks then 2 weeks wash out period followed by 4 weeks for 20 minutes sessions with knee brace (integrated heating pad, a vibration unit and a foot pedal that delivers continuous passive motion)
  Other Names: kineticure system
  Arms: BA

SUMMARY:
The study evaluated the efficacy of combined mechanical vibrations, continuous passive motion and heat on the severity of pain in management of osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OA of the knee by ACR criteria
* symptoms consistent with radiographic OA grades 2, 3 or 4 by Kellgren and Lawrence criteria
* moderate to severe knee pain (≥35mm on a 100mm visual analog pain scale (VAS)).

Exclusion Criteria:

* knee or hip surgery

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
intensity of pain as measured on a 100 mm non-marked VAS and the total Western Ontario McMaster (WOMAC) OA index using a Likert scale, | 10 weeks

SECONDARY OUTCOMES:
satisfaction of use of the Kineticure device as measured on a 0-100 mm non-marked scale | 10 weeks
range of motion (ROM) of the knee (using goniometer) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Kitay, MD, Principal Investigator — Jacksonville Orthopedic Institute
Locations (1):
- Jacksonville Orthopedic Institute, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Kitay GS, Koren MJ, Helfet DL, Parides MK, Markenson JA. Efficacy of combined local mechanical vibrations, continuous passive motion and thermotherapy in the management of osteoarthritis of the knee. Osteoarthritis Cartilage. 2009 Oct;17(10):1269-74. doi: 10.1016/j.joca.2009.04.015. Epub 2009 May 4. PMID 19433134